CLINICAL TRIAL: NCT00655239
Title: Neuroscience-Guided Cognitive Remediation in Adolescents at Risk for Psychosis
Brief Title: Effectiveness of Neuroadaptive Cognitive Training in Adolescents at Risk for Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01MH081051 (NIH); R01MH081051 (NIH)
Record Dates: First submitted 2008-04-07; First posted 2008-04-09 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: Ultra High Risk of Schizophrenia; Prodrome; Psychosis; Schizophrenia; Cognitive Remediation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Participants will use commercially available computer games.
  Interventions: Behavioral: Computer games
- Active (Experimental): Participants will receive targeted neuroadaptive cognitive training with neuroplasticity-based software created by Posit Science Corporation.
  Interventions: Behavioral: Neuroadaptive cognitive training
- Healthy Control (Active Comparator): Healthy participants will receive targeted neuroadaptive cognitive training with neuroplasticity-based software created by Posit Science Corporation.
  Interventions: Behavioral: Neuroadaptive cognitive training

INTERVENTIONS:
Behavioral: Neuroadaptive cognitive training — Neuroadaptive cognitive training includes cognitive remediation exercises that participants will practice 1 hour per day, 5 days per week, for 8 weeks. The exercises are specifically designed to improve speed and accuracy in the perception of and response to verbal targets. The treatment will focus on TCT.
  Arms: Active; Healthy Control
Behavioral: Computer games — The control treatment involves commercially available computer games that participants will practice 1 hour per day, 5 days per week, for 8 weeks.
  Arms: Control

SUMMARY:
This study will evaluate the effectiveness of intensive computerized cognitive training in preventing the onset of psychotic disorder and improving adaptive functioning in adolescents at high risk of schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental disorder that is marked by significant disruption in a person's thought and emotional processes, frequently involving psychotic features. Identifying behavioral changes and symptoms that indicate the beginning stages of schizophrenia is important for early intervention and prevention of a full psychotic episode. These initial symptoms, known as the prodromal symptoms of psychosis, may include odd behaviors, increased social withdrawal, difficulty concentrating, inappropriate emotional responses, suspicion of others, and dramatic sleep and appetite changes. Common treatments for adolescents demonstrating prodromal symptoms include forms of psychotherapy, nutritional training, and low doses of medication. As a form of psychotherapy, neuroadaptive cognitive training exercises delivered on a computer may be the most effective means of remediating the thinking difficulties of adolescents who are experiencing prodromal symptoms and are at risk for developing a first psychotic episode. This study will evaluate the effectiveness of intensive computerized neuroadaptive cognitive training exercises in preventing the onset of psychotic disorder and improving adaptive functioning in adolescents at high risk of schizophrenia.

Participation in this study will last 24 months and will involve both healthy participants and participants at high risk of schizophrenia. Healthy participants will only participate for 12 months. All participants will undergo baseline assessments that will include an interview, written tests, blood draws, and electroencephalogram (EEG) and magnetic resonance imaging (MRI) scans. Participants at high risk of schizophrenia will then be assigned randomly to receive treatment with either computerized neuroadaptive cognitive training or commercially available computer games. Healthy participants will receive treatment with computerized neuroadaptive cognitive training only. All participants will be asked to complete 60-minute sessions of their assigned treatments 5 days per week for 8 weeks. For participants receiving cognitive training, exercises will focus on improving speed and accuracy in the perception of and response to verbal and visuospatial targets. The treatment will focus on targeted cognitive training (TCT). Participants assigned to practice computer games will play standard, commercially available games, with no targeted response.

Participants will repeat baseline assessments at post treatment and Month 6 of follow-up. The EEG and MRI will be repeated only at the Week 8 assessment visit. There will be a blood draw at Week 2 of treatment as well. After the Month 6 assessment, healthy controls will be complete, and the at risk participants will continue to be followed up out to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria from the Structured Interview of Prodromal Syndromes for the diagnosis of a prodromal syndrome
* Good general physical health
* English is first language
* Clinically stable (e.g., outpatient status for at least 8 weeks before study entry;on stable doses of medications for at least 1 month before study entry)

Exclusion Criteria:

* Confirmed neurological disorder

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2008-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cognitive performance, as measured by a neuropsychological battery | Measured at baseline, Weeks 8 and Month 6, 12, 18, and 24 follow-up

SECONDARY OUTCOMES:
Symptom profile, as measured by clinical interviews | Measured at baseline, Weeks 8 and Month 6, 12, 18, and 24 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of California, San Francisco; San Francisco VA Medical Center; NCIRE - The Veterans Health Research Institute; Rachel Loewy, PhD, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Loewy R, Fisher M, Schlosser DA, Biagianti B, Stuart B, Mathalon DH, Vinogradov S. Intensive Auditory Cognitive Training Improves Verbal Memory in Adolescents and Young Adults at Clinical High Risk for Psychosis. Schizophr Bull. 2016 Jul;42 Suppl 1(Suppl 1):S118-26. doi: 10.1093/schbul/sbw009. Epub 2016 Feb 22. PMID 26903238